CLINICAL TRIAL: NCT04734860
Title: A Randomized, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Efficacy of a Single Dose of STI-2020 (COVI-AMG™) in Adults With Mild COVID-19 Symptoms
Brief Title: Study to Evaluate a Single Dose of STI-2020 (COVI-AMG™) in Adults With Mild COVID-19 Symptoms
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A different study will be conducted.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMG-COV-201
Record Dates: First submitted 2021-01-29; First posted 2021-02-02 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-AMG (Experimental): A single injection of 40 mg, 100 mg, or 200 mg of COVI-AMG will be administered
  Interventions: Biological: COVI-AMG
- Placebo (Placebo Comparator): A single injection of placebo will be administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-AMG — COVI-AMG is a fully human SARS-CoV-2 neutralizing monoclonal antibody (mAb)
  Other Names: STI-2020
  Arms: COVI-AMG
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This study investigates the safety, pharmacokinetic (PK) profile and efficacy of a single injection of COVI-AMG in outpatient adults with mild COVID-19 symptoms.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind study designed to investigate the safety, pharmacokinetic (PK) profile and efficacy of a single injection of COVI-AMG in outpatient adults with mild COVID-19 symptoms. Subjects will be followed for approximately 70 days post dosing.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID-19 by an approved antigen test
* Mild symptoms consistent with a COVID-19 viral infection
* Willing and able to comply with all planned study procedures and be available for all study visits and follow-up as required by the protocol
* Willing to follow contraception guidelines

Exclusion Criteria:

* Evidence of moderate COVID-19 per FDA severity categorization
* Pregnant or lactating and breast feeding or planning on either during the study
* Has a documented infection other than COVID-19
* Has received a COVID-19 vaccine
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies (mAbs) against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who have remained out of the hospital or emergency room through Day 29 | Randomization to Day 29
  Proportion of subjects who have remained out of the hospital or emergency room through Day 29

SECONDARY OUTCOMES:
Viral load reduction from baseline to Day 8, 15, 29, 43, and 70 | Randomization to Day 8, 15, 29, 43, 70
  Viral load reduction from baseline to Day 8, 15, 29, 43, and 70 as assessed by nasopharyngeal RT-PCR test
Proportion of subjects who have remained out of the hospital or emergency room through Day 43 and 70 | Randomization to Day 43 and Day 70
  Proportion of subjects who have remained out of the hospital or emergency room through Day 43 and 70
Proportion of subjects who have 50%, 70%, and 90% reduction in PRO instrument score | Randomization to Day 15, 29, 43
  Proportion of subjects who have 50%, 70%, and 90% reduction in PRO instrument score from baseline at Day 15, 29, and 43
Time to resolution of fever | Randomization through study completion at Day 70
  For subjects who have a fever at randomization, time to resolution of the fever

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics
Locations (4):
- United States (4):
  - Collaborative NeuroScience Research, LLC, Garden Grove, California
  - Synergy Healthcare LLC, Bradenton, Florida
  - Med-Care Research, Miami, Florida
  - ETNA Medical Center, Tamarac, Florida

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343